CLINICAL TRIAL: NCT04360044
Title: Efficacy of Inhaled Cannabis Versus Placebo for the Acute Treatment of Migraine: a Randomized, Double-blind, Placebo-controlled, Crossover Trial
Brief Title: Efficacy of Inhaled Cannabis for Acute Migraine Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Migraine Research Foundation (Other)
Responsible Party: Principal Investigator, Nathaniel Schuster, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018 MRF Impact Award
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Migraine; Cannabis; THC; CBD
Keywords: Migraine; Cannabis; THC; CBD
MeSH Terms: conditions — Migraine Disorders; Marijuana Abuse | interventions — THC 5; Dronabinol; nabiximols; Cannabidiol; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blind, Placebo-controlled, Crossover Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Each participant will have an identification number and randomization of drug sequence allocation will be performed a priori using a random number generator by the study pharmacist. The 4 treatments will be identically encapsulated by the study pharmacist using Storz & Bickel filling set. The study pharmacist will place the capsules in identical sealed plastic bags labeled "Migraine 1" through "Migraine 4."
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- THC ~5% (Experimental): 4 puffs of cannabis flower containing THC ~5% administered by vaporizer using Foltin Uniform Puff Procedure for treatment of a moderate-severe migraine attack. The flower is from the United States National Institute on Drug Abuse (NIDA).
  Interventions: Drug: THC ~5%
- THC ~5%/CBD ~12% (Experimental): 4 puffs of cannabis flower containing THC ~5% and CBD ~12% administered by vaporizer using Foltin Uniform Puff Procedure for treatment of a moderate-severe migraine attack. The flower is from the United States National Institute on Drug Abuse (NIDA).
  Interventions: Drug: THC ~5% and CBD ~12%
- CBD ~12% (Experimental): 4 puffs of cannabis flower containing CBD ~12% administered by vaporizer using Foltin Uniform Puff Procedure for treatment of a moderate-severe migraine attack. The flower is from the United States National Institute on Drug Abuse (NIDA).
  Interventions: Drug: CBD ~12%
- Sham Cannabis (Sham Comparator): 4 puffs of cannabis flower from which the THC and CBD have been extracted administered by vaporizer using Foltin Uniform Puff Procedure for treatment of a moderate-severe migraine attack. The flower is from the United States National Institute on Drug Abuse (NIDA).
  Interventions: Drug: Sham Cannabis

INTERVENTIONS:
Drug: THC ~5% — 4 puffs of vaporized flower containing THC ~5%
  Other Names: THC; delta 9-tetrahydrocannabinol; marijuana
  Arms: THC ~5%
Drug: CBD ~12% — 4 puffs of vaporized flower containing CBD ~12%
  Other Names: CBD; cannabidiol; hemp
  Arms: CBD ~12%
Drug: THC ~5% and CBD ~12% — 4 puffs of vaporized flower containing THC ~5% and CBD ~12%
  Other Names: THC; CBD; delta 9-tetrahydrocannabinol; cannabidiol; marijuana; hemp
  Arms: THC ~5%/CBD ~12%
Drug: Sham Cannabis — 4 puffs of vaporized flower from which the THC and CBD have been extracted
  Other Names: Placebo; Sham
  Arms: Sham Cannabis

SUMMARY:
This crossover study will evaluate 3 different treatments of vaporized cannabis (THC, THC/CBD mix, and CBD) and vaporized placebo cannabis for the acute treatment of migraine.

DETAILED DESCRIPTION:
In this double-blind, randomized, crossover trial, subjects will treat 4 separate migraine attacks with 4 different treatments. Inhaled cannabis will be administered using a portable vaporization system (Mighty Medic; Storz & Bickel) based on a validated Storz & Bickel system and using a standardized inhalation approach. Subjects will self-administer inhaled cannabis as early as possible in the course of a migraine (see Procedure), taking 4 puffs of 1) THC, 2) THC/CBD mix, 3) CBD, or 4) placebo. Patients will treat each of the 4 distinct migraine attacks with a different cannabis sample. Outcomes measured will include pain freedom and pain relief as well as presence or absence of photophobia, phonophobia, and nausea at 1 hour, 2 hours (primary outcome), 24 hours, and 48 hours.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 21 and ≤ 65
* Able to communicate in English
* Migraine, with or without aura, in its episodic or chronic manifestations, as per the International Headache Society (IHS) classification International Classification of Headache Disorders (ICHD-3) criteria (section 1.1, 1.2, 1.3).(48)
* Ability to provide informed consent and complete website questionnaires in English
* Agrees not to use cannabis outside of the study during participation in the study
* Agrees not to use opioids or barbiturates during participation in the study
* Agrees not to drive a motor vehicle within 4 hours following last use of inhaled cannabis during participation in the study

Exclusion Criteria:

* Positive urine drug test for THC, barbiturates, opioids, oxycodone, or methadone prior to enrollment
* Pregnancy
* Breastfeeding
* Prisoner
* Known cognitive impairment
* Institutionalized
* Current moderate-severe or severe depression
* Current or past history of bipolar depression, schizophrenia, or psychosis
* Current or past history of cannabis, alcohol, opioid, or amphetamine abuse or other substance use disorder at the discretion of the research team
* Active pulmonary disease class IV heart failure, cirrhosis, or other severe medical illnesses at the discretion of the research team.
* Allergy or past adverse effects or negative past experiences from cannabis

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Headache Pain Relief at 2 Hours Post-Treatment | 2 Hours Post-Treatment
  Dichotomous endpoint of pain reduction defined as reduction from moderate/severe pain to mild/no pain

SECONDARY OUTCOMES:
Headache pain freedom | 2 hours
  Dichotomous endpoint of reduction from moderate/severe pain to no pain
Most bothersome symptom freedom | 2 hours
  Dichotomous endpoint of resolution of most bothersome symptom (of photophobia, phonophobia, and nausea) selected at the beginning of the migraine prior to cannabis administration

OTHER OUTCOMES:
Headache pain relief | 1 hour, 24 hours, 48 hours
  Dichotomous endpoint of reduction from moderate/severe pain to mild/no pain
Headache pain freedom | 1 hour, 24 hours, 48 hours
  Dichotomous endpoint of reduction from moderate/severe pain to no pain
Most bothersome symptom freedom | 1 hour, 24 hours, 48 hours
  Dichotomous endpoint of resolution of most bothersome symptom (of photophobia, phonophobia, and nausea) selected at the beginning of the migraine prior to cannabis administration
Freedom from photophobia | 1 hour, 2 hours, 24 hours, 48 hours
  Dichotomous endpoint of resolution of photophobia
Freedom from phonophobia | 1 hour, 2 hours, 24 hours, 48 hours
  Dichotomous endpoint of resolution of phonophobia
Freedom from nausea | 1 hour, 2 hours, 24 hours, 48 hours
  Dichotomous endpoint of resolution of nausea
Freedom from vomiting | At any time over 48 hours
  Dichotomous endpoint of whether patient vomited during this migraine attack
Use of rescue medication | At any time over 48 hours
  Dichotomous endpoint of use of rescue medication
Sustained pain freedom | 24 hours and 48 hours
  Dichotomous endpoint of absence of headache pain at 2 hours after dose, with no use of rescue medication and no relapse of headache pain
Sustained most bothersome symptom freedom | 24 hours and 48 hours
  Dichotomous endpoint of absence of most bothersome symptom at 2 hours afer dose, with no use of rescue medication and no relapse of most bothersome symptom

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel M Schuster, MD, Principal Investigator — University of California, San Diego
Locations (1):
- Center for Pain Medicine, UC San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared in a manner TBD based on funding availability and journal requirements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 1 year and ending 5 years after article publication
Access Criteria: Researchers who provide a methodologically sound proposal. Proposals should be sent to nmschuster@health.ucsd.edu.